CLINICAL TRIAL: NCT07310056
Title: The Construction and Clinical Application of an Integrated Perioperative Management System for Lung Cancer Based on Wearable Devices and Intelligent Platforms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xuelei Ma MD, Department of Biotherapy, West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Approval No. 1647 (2024)
Record Dates: First submitted 2025-11-30; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Rehabilitation; Thoracic Surgery; Perioperative Management
Keywords: Non-Small Cell Lung Cancer; Lung Cancer Surgery; Wearable Devices; Perioperative Management; Rehabilitation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients in this arm receive standard perioperative care plus a wearable-based digital perioperative rehabilitation program. The intervention includes preoperative personalized exercise training (aerobic exercise, respiratory muscle training, and resistance training), real-time six-minute walk test monitoring, portable pulmonary function testing, and continuous physiological monitoring using wearable devices (heart rate, oxygen saturation, and activity level). After discharge, patients undergo a 30-day home-based digital rehabilitation program with daily exercise tasks, real-time data upload, electronic patient-reported outcomes (ePROs), and remote guidance via a digital platform. Rehabilitation plans are dynamically adjusted based on patient performance and physiological data.
  Interventions: Device: Wearable-Based Digital Perioperative Rehabilitation System
- Standard Perioperative Care (Active Comparator): Patients in this arm receive standard perioperative management only. This includes routine preoperative assessment, standardized surgical and anesthesia care, and conventional postoperative rehabilitation guidance at discharge. No wearable device monitoring, prehabilitation training, or digital home-based rehabilitation platform is provided. Patients are followed according to routine outpatient follow-up schedules after discharge.
  Interventions: Behavioral: Standard Perioperative Rehabilitation Guidance

INTERVENTIONS:
Device: Wearable-Based Digital Perioperative Rehabilitation System — This intervention consists of a wearable-based digital perioperative rehabilitation system designed for patients with non-small cell lung cancer undergoing thoracic surgery. The system integrates continuous physiological monitoring, functional assessment, and remote rehabilitation management. During the preoperative phase, patients receive personalized prehabilitation including aerobic exercise, respiratory muscle training, and resistance training. Wearable devices continuously monitor heart rate, oxygen saturation, activity level, and walking distance, including real-time monitoring during the six-minute walk test. Portable pulmonary function testing and functional MRI (PREFUL) are used for baseline assessment. During the postoperative phase, patients receive 30 days of home-based digital rehabilitation, including daily exercise tasks, real-time data upload, electronic patient-reported outcomes, and remote feedback from clinicians via a digital platform. Rehabilitation plans are dynam
  Arms: Experimental
Behavioral: Standard Perioperative Rehabilitation Guidance — This behavioral intervention consists of standard perioperative rehabilitation guidance provided to patients undergoing thoracic surgery for non-small cell lung cancer. Patients receive routine preoperative assessment, standardized postoperative discharge education, and conventional rehabilitation instructions including breathing exercises, early mobilization, pain management, and activity recommendations. No structured prehabilitation program, wearable device monitoring, remote digital platform, or continuous physiological monitoring is provided. Post-discharge follow-up is conducted according to routine outpatient clinical practice.
  Arms: Standard Perioperative Care

SUMMARY:
This study aims to develop and evaluate an integrated perioperative management system based on wearable devices and a digital rehabilitation platform for patients with non-small cell lung cancer (NSCLC) undergoing thoracic surgery. By combining preoperative functional assessment using the six-minute walk test (6MWT), continuous perioperative physiological monitoring, and structured postoperative home-based digital rehabilitation, this randomized controlled trial will investigate whether the wearable-based digital management model improves short-term postoperative pulmonary function, functional recovery, and clinical outcomes compared with standard perioperative care.

DETAILED DESCRIPTION:
With the rapid development of wearable sensor technology and digital health platforms, continuous physiological monitoring and remote rehabilitation have become feasible throughout the perioperative period. However, current perioperative management for lung cancer patients remains fragmented, with limited integration of preoperative functional assessment, intraoperative monitoring, and postoperative home-based rehabilitation. This study is designed to establish and validate a comprehensive wearable-based perioperative management system for patients with non-small cell lung cancer (NSCLC) undergoing surgical resection.

This study is a prospective, single-center, randomized, single-blind, superiority-controlled trial. A total of 126 eligible patients undergoing elective video-assisted thoracoscopic lobectomy or segmentectomy will be randomly assigned in a 1:1 ratio to either the intervention group or the control group. The control group will receive standard perioperative management and routine postoperative rehabilitation guidance. The intervention group will receive standard care plus a digital perioperative rehabilitation program supported by wearable devices and a remote monitoring platform.

During the preoperative phase, patients in the intervention group will undergo personalized prehabilitation including aerobic exercise training, respiratory muscle training, and resistance exercise. The six-minute walk test (6MWT), portable pulmonary function testing, and non-contrast functional lung MRI (PREFUL technology) will be performed for functional assessment. Wearable devices will continuously collect heart rate, blood oxygen saturation, step count, and activity level.

During the intraoperative phase, standardized surgical procedures and anesthetic management will be applied. Key intraoperative indicators including blood loss, ventilation time, anesthesia duration, and complications will be recorded through the anesthesia and surgical information systems.

During the postoperative phase, patients in the intervention group will receive 30-day home-based digital rehabilitation, including daily exercise tasks, real-time wearable data upload, electronic patient-reported outcomes (ePROs) reporting of symptoms (pain, fatigue, dyspnea), and remote review and guidance by medical staff via the digital platform. The control group will receive routine discharge education and outpatient follow-up.

The primary endpoint of the study is the between-group difference in pulmonary function (FEV₁, FVC, FEV₁/FVC) at 30 days and 3 months after surgery. Secondary endpoints include six-minute walk distance, peak oxygen consumption (VO₂ peak), postoperative complications, chest tube duration, length of hospital stay, time to first ambulation, 30-day readmission rate, analgesic consumption, symptom burden assessed using the MD Anderson Symptom Inventory-Lung Cancer module (MDASI-LC), and rehabilitation adherence based on platform usage data.

By integrating wearable-based continuous monitoring, objective functional assessment, and structured digital rehabilitation, this study aims to establish a closed-loop, data-driven perioperative management model. The results are expected to provide high-quality clinical evidence for the effectiveness, safety, and feasibility of wearable-assisted perioperative rehabilitation in lung cancer patients, and to promote the clinical translation of digital health technologies into thoracic surgery practice.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years and ≤85 years

Pathologically confirmed primary non-small cell lung cancer (NSCLC)

Scheduled to undergo elective curative-intent thoracoscopic lobectomy or segmentectomy

Postoperative clinical condition is stable and judged by investigators to be suitable for discharge within 2-7 days after surgery

Able to independently operate a smartphone and wearable device, or able to do so with caregiver assistance

Willing to comply with study procedures and follow-up requirements

Provided written informed consent prior to participation

Exclusion Criteria:

Preoperative long-term home oxygen therapy or severe resting respiratory failure

Presence of severe or uncontrolled cardiopulmonary disease, cerebrovascular disease, hepatic insufficiency, or renal insufficiency

Severe comorbid conditions that significantly limit physical activity or adherence to rehabilitation

Known or suspected allergy to materials used in wearable devices or medical adhesives

Severe postoperative complications requiring reoperation or prolonged mechanical ventilation

Occurrence of serious adverse events during the six-minute walk test that prevent continuation of the study

Any other condition that, in the judgment of the investigators, makes the participant unsuitable for study participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in 1 Second (FEV₁) | Baseline (preoperative), 30 days after surgery, and 3 months after surgery
  Change in forced expiratory volume in 1 second (FEV₁), measured by spirometry, comparing postoperative pulmonary function recovery between the wearable-based digital rehabilitation group and the standard care group. Unit of Measure: Liters (L)

SECONDARY OUTCOMES:
Six-Minute Walk Distance (6MWD) | Baseline (preoperative), 30 days after surgery, and 3 months after surgery
  The change in six-minute walk distance will be used to evaluate functional exercise capacity and recovery after surgery.
Change in Forced Vital Capacity (FVC) | Baseline (preoperative), 30 days after surgery, and 3 months after surgery
  Change in forced vital capacity (FVC), measured by spirometry, comparing postoperative pulmonary function recovery between the wearable-based digital rehabilitation group and the standard care group.
Change in FEV₁/FVC Ratio | Baseline (preoperative), 30 days after surgery, and 3 months after surgery
  Change in the ratio of forced expiratory volume in 1 second to forced vital capacity (FEV₁/FVC), measured by spirometry, comparing postoperative pulmonary function recovery between the wearable-based digital rehabilitation group and the standard care group.
Peak Oxygen Consumption (VO₂ peak) | 30 days and 3 months after surgery
  Peak oxygen consumption measured by cardiopulmonary exercise testing will be used to assess cardiorespiratory fitness.
Postoperative Complication Rate | From surgery to 30 days after surgery
  The incidence of postoperative complications including pulmonary infection, atelectasis, prolonged air leak, pain, postoperative nausea and vomiting, and venous thromboembolism.
Length of Postoperative Hospital Stay | From the date of surgery until the date of hospital discharge, assessed up to 90 days after surgery.
  Total number of days of hospitalization after surgery.
Quality of Life (MDASI-LC) | Baseline (preoperative), 30 days after surgery, and 3 months after surgery
  Quality of life and symptom burden will be assessed using the MD Anderson Symptom Inventory-Lung Cancer module (MDASI-LC), which evaluates pain, fatigue, dyspnea, sleep disturbance, and overall symptom severity in patients with lung cancer.

OTHER OUTCOMES:
Regional Lung Function by Functional MRI (PREFUL) | Baseline (preoperative), 1 and 3 months after surgery
  Regional ventilation and perfusion parameters evaluated by non-contrast functional MRI to assess postoperative regional lung function recovery.